CLINICAL TRIAL: NCT02944968
Title: Clinical Study for Workflow and Acute Performance Evaluation of the THERMOCOOL SMARTTOUCH® SF-5D System (the THERMOCOOL SMARTTOUCH® SF-5D Catheter With Temperature Sensing Capabilities and Micro Electrodes and CARTO 3 V 6.0 Technology) in Treatment of Patients With Paroxysmal Atrial Fibrillation (QDOT-Micro)
Brief Title: Clinical Study for Workflow and Performance Evaluation of the THERMOCOOL SMARTTOUCH® SF-5D System for Treating Symptomatic Paroxysmal AF (QDOT-Micro)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MQDT-166
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Interventional; Radiofrequency Ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment group (Experimental): Radiofrequency ablation treatment with the THERMOCOOL SMARTTOUCH® SF-5D catheter in Paroxysmal AF population.
  Interventions: Device: THERMOCOOL SMARTTOUCH® SF-5D catheter

INTERVENTIONS:
Device: THERMOCOOL SMARTTOUCH® SF-5D catheter

SUMMARY:
The QDOT-Micro study is a prospective, multi-center, non-randomized, interventional clinical study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the workflow and acute performance , during standard electrophysiology mapping and RF ablation procedures, of the THERMOCOOL SMARTTOUCH® SF-5D catheter with temperature sensing capabilities and micro electrodes used in combination with the CARTO® 3 Navigation System with THERMOCOOL SMARTTOUCH® SF-5D-module.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following criteria:

1. Age 18 or older
2. Patients who have signed the Patient Informed Consent Form (ICF)
3. Subjects diagnosed with symptomatic documented PAF* who are candidates for catheter ablation
4. Able and willing to comply with all pre-, post-, and follow-up testing and requirements (eg. Patient not confined by a court ruling)

Exclusion Criteria:

Candidates for this study will be EXCLUDED from the study if ANY of the following conditions apply:

1. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Previous ablation for atrial fibrillation.
3. Previously diagnosed with persistent AF.
4. Documented Left Atrial thrombus
5. Any carotid stenting or endarterectomy
6. LA size >50mm
7. LVEF <40%
8. Uncontrolled heart failure or NYHA function class III and IV
9. History of blood clotting or bleeding abnormalities or contraindication to anticoagulation ( heparin, warfarin, or dabigatran)
10. History of a documented thromboembolic event (including TIA) within the past 12 months.
11. Previous PCI/MI within the past 3 months
12. Previous cardiac surgery (e.g CABG) in conjunction with valve surgery or any valvular cardiac surgical/percutaneous procedure (e.g ventriculotomy, atriomy, valve repair or replacement, presence of a prosthetic valve) within the past 6 months.
13. Awaiting cardiac transplantation or other cardiac surgery within the next 6 months.
14. Unstable angina
15. Significant pulmonary disease (eg, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
16. Acute illness, active systemic infection, or sepsis.
17. Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation.
18. Presence of a condition that precludes vascular access.
19. Presence of implantable cardioverter-defibrillator (ICD)
20. Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this trial.
21. Currently enrolled in an investigational study evaluating another device, biologics, or drug.
22. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the clinical investigation (as evidenced by pregnancy test if of child bearing potential).
23. Life expectancy less than 12 months.
24. Presenting contra-indication for the devices used in the study, as indicated in the respective instructions for use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 subjects were enrolled in the study at 6 sites in Europe. The first subject was enrolled on September 28th, 2016 and the last subject was enrolled on April 26th, 2018.
Pre-assignment Details: Subjects were screened carefully prior to enrollment in the study to ensure compliance with the inclusion and exclusion criteria. All subjects had pre-procedure imaging to screen for the presence of left atrial appendage thrombus to decrease the potential for thromboembolic complications.
Groups:
- THERMOCOOL SMARTTOUCH® SF-5D: The THERMOCOOL SMARTTOUCH® SF-5D Catheter with improved temperature sensing capabilities and micro electrodes and CARTO®3 V6 technology
Period: Overall Study
Arm/Group | THERMOCOOL SMARTTOUCH® SF-5D
Started (Enrolled subjects (under protocol v1.0 and v2.0).) | 51
Completed (Evaluable subjects (under protocol v1.0 and v2.0) who completed the study.) | 48
Not Completed | 3
Not completed — Subject excluded before study procedure | 1
Not completed — Subject didn't meet eligibility criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | THERMOCOOL SMARTTOUCH® SF-5D
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  European Union | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Entrance Block Confirmation in the Total Effectiveness Outcome Population
Description: Confirmation of entrance block in all targeted PVs after adenosine and/or isoproterenol challenge achieved at the end of procedure. If the challenge was not done, confirmation data would not be available.
Time Frame: Day of ablation procedure
Population: This total effectiveness outcome population includes all subjects (under both protocols v1.0 and v2.0), complied with study inclusion and exclusion criteria, received investigational device, and had an adenosine challenge applied for verifying entrance block.
Measure: Count of Participants; unit: Participants
Arm/Group | THERMOCOOL SMARTTOUCH® SF-5D
Number analyzed (Participants) | 47
Participants
  Subjects with entrance block confirmation | 46
  Subjects without entrance block confirmation | 1

2. Secondary Outcome: Number of Participants With Early Onset Primary Adverse Events in Total Safety Population
Description: Primary adverse events include Death, Atrio-Esophageal Fistula, Cardiac Tamponade/Perforation, Myocardial Infarction, Stroke/Cerebrovascular Accident, Thromboembolism, Transient Ischemic Attack, Diaphragmatic Paralysis, Pneumothorax, Heart Block, Pulmonary Vein Stenosis, Pulmonary Edema (Respiratory Insufficiency), Vagal Nerve Injury, Pericarditis, Major Vascular Access Complication/Bleeding, Pulmonary vein (PV) stenosis and atrio-esophageal fistula
Time Frame: Seven Days Post Procedure
Population: Total Safety Population: includes subjects enrolled under CIP v1.0 and 2.0 who underwent study procedure with investigational device.
Measure: Count of Participants; unit: Participants
Arm/Group | THERMOCOOL SMARTTOUCH® SF-5D
Number analyzed (Participants) | 50
Participants
  Subjects with Pericard. effusion without tamponade | 1
  Subjects with Pericarditis | 1
  Subjects with Vascular pseudoaneurysm | 1
  Subjects without primary adverse events | 47

ADVERSE EVENTS:
Time Frame: Three months follow up after procedure
Description: An AE is any untoward medical occurrence/clinical sign/unintended disease/injury in subjects/users/other persons, related or not to the investigational device.
Arm/Group | THERMOCOOL SMARTTOUCH® SF-5D
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 7/50
Other Adverse Events (participants affected / at risk) | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL SMARTTOUCH® SF-5D (N=50)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL SMARTTOUCH® SF-5D (N=50)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Thyroid disorder (Endocrine disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 6 (6)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haematoma (Vascular disorders) | 5 (5)
Perforation (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.

DOCUMENTS (2):
  • Study Protocol (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT02944968/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02944968/SAP_001.pdf